CLINICAL TRIAL: NCT04778813
Title: Evaluation of Three Artemisinin-based Combinations for the Treatment of Uncomplicated Malaria in Childreen in Burkina Faso (CHIMIO2)
Acronym: CHIMIO2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre national de recherche et de formation sur le paludisme (Other Government)
Collaborators: Programme national de lutte contre le paludisme (PNLP), Burkina Faso (Unknown); Unité de recherche clinique de Nanoro (URCN) (Unknown); USAID/IMPACT Malaria (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TET2020_001
Record Dates: First submitted 2021-02-24; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Malaria; Burkina Faso
Keywords: Plasmodium falciparum; Treatment; ACT; Childreen
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination; pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, open-label, three-arm study involving three sites representing the three different epidemiological facies of malaria in Burkina Faso.The three therapeutic combinations (AL, DHA-PPQ and As-Pyr) will be tested in different sites with different characteristics of transmission and resistance of malaria. Participants will be treated for 3 days then followed during by 28-days (AL arm) and 42-days (DHA-PPQ and Pas-Pyr). There will be no comparision between study arms, but the for each arm, the efficacy will be measured and compared to WHO critical value.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Artemether-lumefantrin (AL) (Experimental): The tablets will be given orally according to patients' age and under supervision of study team as follows:
  * Day 0: H0 and H8
  * Day 1: H24 and H36
  * Day 2: H48 and H60
  Interventions: Drug: Artemether-lumefantrine
- Dihydro-artemisinin-piperaquin (DHA-PPQ) (Experimental): The tablets will be given orally according to patients' age and under supervision of study team as follows. A single dose will be given on day 0, 1 and 2
  Interventions: Drug: Artemether-lumefantrine
- Artesunate-Pyronaridin (As-Pyr) (Experimental): The tablets will be given orally according to patients' age and under supervision of study team as follows. A single dose will be given on day 0, 1 and 2
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Artemether-lumefantrine — In each study site, children fulfilling the inclusion criteria will be assigned randomly to one of three treatment groups: AL, DHA-PPQ or As-Pyr group. Sealed envelopes each containing no more than 10 other small envelopes with randomization numbers and treatment will also be provided. These will be used over time, respecting the ascending order of the numbers to randomly distribute the eligible children after selection in each of the three treatment groups. The treatment to be administered will not be known until after the randomization process. The drugs will be administered based on weight according to the instructions from the drug manufacturer. AL will be administered with fatty food or milk according to the manufacturer's recommendations. All doses of the drug will be administered under the direct supervision of a qualified team member designated by the principal investigator.
  Other Names: Dihydroartemisinin pyperaquin; Artesunate Pyronaridine

SUMMARY:
Bakground In Burkina Faso, since the adoption of this new malaria treatment policy in 2005, several studies evaluating the efficacy and tolerance of ACTs have been carried out by different research teams at different sites according to an irregular chronology and according to different methods. Studies conducted in children 6 to 59 months with supervised use of ACTs indicate adequate clinical and parasitological response rates varying between 93% to 98% after correction to the PCR at day 28. With the introduction of seasonal malaria chemoprevention (SMC) by the Sulfadoxine-Pyriméthamime/amodiaquine combination in almost all health districts of Burkina Faso, ASAQ is no longer recommended for the treatment of uncomplicated malaria in the areas covered by this intervention. In 2017, DHA-PPQ was added to the national treatment guidelines as a first-line treatment option. The therapeutic efficacy study carried out in 2017-2018 by the CNRFP showed a PCR-corrected treatment failure rate of over 10% with the AL combination. However, molecular analyzes have not shown the presence of mutations at position 580 on the PfK-13 gene which is associated with resistance to artemisinin derivatives. The combination artesunate-pyronaridine (As-Pyr) was recently added to the WHO Prequalified Medicines List and Essential Medicines List. In 2019, it received regulatory marketing authorization to be used as a treatment for malaria in Burkina Faso. Burkina Faso (along with the Niangoloko and Bobo Dioulasso centers) was one of the countries where clinical trials p ar the As-Pyr association were led. This combination has been found to be effective and well tolerated in Burkina Faso. The combinations of AL and DHA-PPQ were observed to be well tolerated in previous efficacy studies. The combinations DHA-PPQ and As-Pyr could potentially replace AL as first-line treatment in Burkina Faso if the results of these planned therapeutic efficacy studies continue to show a high rate of failures with AL. The herein study aims to assess the efficacy and safety of AL, DHA-PPQ and As-Pyr in the treatment of uncomplicated malaria in children in three health districts in Burkina Faso, namely the health districts of Banfora, Nanoro and de Gourcy. This study will provide PNLP and the Ministry of Health with additional data and evidence on the safety and efficacy of these treatments against malaria in Burkina Faso.

Primary objective The primary objective is to assess the clinical and parasitological efficacy of AL, DHA-PPQ and AS-Pyr in the treatment of uncomplicated P. falciparum malaria in children aged 6 months to 12 years, corrected by PCR on day 28 (AL) or 42 (DHA-PPQ & AS-Pyr).

Study settings The study will be conducted at the medical center (CMA of Niangoloko, the Clinical Research Unit of Nanoro (URCN) and the medical center with surgical antenna (CMA) of Gourcy.

Populations Febrile patients of both sexes aged between 6 months and 12 years with confirmed uncomplicated P. falciparum mono-infestation who wellcome for an outpatient visit to the health facilities.

Procedures It will be a multicenter, randomized, open-label, three-arm study involving three sites representing the three epidemiological facies of malaria in Burkina Faso. The three therapeutic combinations (AL, DHA-PPQ and As-Pyr) will be tested in different sites with different characteristics of transmission and resistance of malaria. Children with uncomplicated malaria who meet the criteria for inclusion in the study will be recruited and treated with the combination of AL or DHA-PPQ or As-Pyr. They will be monitored for 28 days for the AL group and 42 days for the DHA-PPQ and AS-Pyr arm. The follow-up will consist of scheduled control visits during which clinical examinations and laboratory tests will be carried out. A total of 1050 children will be enrolled in the study.

Main results

1. The proportion of patients with early treatment failure, late clinical failure, late parasitological failure or adequate clinical and parasitological response.
2. The frequency and nature of adverse events.
3. The blood concentration of lumefantrine on day 7

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes aged 6 months to 12 years inclusive;
* Microscopic confirmation of a monospecific infection by P. falciparum (Parasitaemia between 2000 - 200,000 / μl);
* Fever (uncorrected axillary or tympanic temperature ≥37.5 ° C or history of fever reported within the last 24 hours
* Hemoglobin level ≥ 5.0 g / dl
* Ability to take oral medication;
* Ability and willingness of parents to respect the protocol for the duration of the study and to respect the consultation schedule;
* Signature (or fingerprint (thumb) when parents / guardians are illiterate) of the consent form by the child's parents or guardians.

Exclusion Criteria:

* General danger signs in children under five (inability to drink or breastfeed, repeated vomiting (> 2 times in 24 hours), convulsions, unconsciousness, inability to sit or stand standing)
* Body weight less than 5 kg;
* Fever due to illnesses other than malaria (e.g. measles, acute lower respiratory infection, severe diarrheal illness with dehydration) or presence of other known chronic or serious underlying illnesses or any other condition (e.g. illness cardiac, renal or hepatic, HIV / AIDS) which in the judgment of the clinical investigator would place the subject at potential risk or interfere with the conduct of the study;
* Previous complete antimalarial treatment with an ACT within the last two weeks;
* History of hypersensitivity to any of the drugs tested
* Severe malnutrition (defined by a z score of weight for age less than -3 or other severe malnutrition sign).
* Known individual or family history of clinical disorders of prolongation of QT intervals or sudden death
* Previous participation in a malaria vaccine clinical trial

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1050 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Early treatment failure | 3 days
  * danger signs or severe malaria on Day 1, 2, or 3 in the presence of parasitemia;
  * parasite count on Day 2 higher than on Day 0, irrespective of axillary temperature;
  * parasitemia on Day 3 with axillary temperature ≥37.5°C;
  * parasite count on Day 3 ≥25% on Day 0
Late clinical failure | 24 days
  * danger signs or severe malaria on any day between Day 4 and Day 28 in the presence of parasitemia, without previously meeting any of the criteria of early treatment failure;
  * presence of parasitemia and axillary temperature ≥37.5°C (or history of fever) on any day between Day 4 and Day 28, without previously meeting any of the criteria of early treatment failure
Late parasitological failure | 21 days
  Presence of parasitemia on any day between Day 7 and Day 28 and axillary temperature <37.5°C, without previously meeting any of the criteria of early treatment failure or late clinical failure.
Day 28 Adequate clinical and parasitological response PCR corrected | 28 days
  Absence of parasitaemia by day 28 without previously meeting any of the criteria for ETF, LCF and LPF. The number of cases of total treatment failure (TTF) will be computed as ETF+LCF+LPF

SECONDARY OUTCOMES:
Adverse events frequency and type | 28 days
  Any unwanted sign/symptom occurred in patients after consentement signature
Pharmacocinetic of Lumefantrin | 7 days
  Concentration of lumefantrin in blood at day 7 after IP administration

CONTACTS AND LOCATIONS:
Overall Officials: Adama Gansane, PhD, Principal Investigator — Centre national de recherche et de formation sur le paludisme
Locations (1):
- Centre national de recherche et de formation sur le paludisme (CNRFP), Ouagadougou, Kadiogo, Burkina Faso